CLINICAL TRIAL: NCT03627793
Title: Resistance Exercise Training at Different Intensities in Healthy and Frail Older People: A Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Glasgow (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Principal Investigator, Dr Evan Campbell, Research Associate, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3.0
Record Dates: First submitted 2018-08-02; First posted 2018-08-13 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Frail Elderly Syndrome
Keywords: frailty; exercise; resistance training; strength; older adults
MeSH Terms: conditions — Frailty; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High load non-frail (Active Comparator): Non-frail participants who will receive resistance training at 70% of their maximal strength
  Interventions: Other: resistance training
- low load non-frail (Active Comparator): Non-frail participants who will receive resistance training at 30% of their maximal strength
  Interventions: Other: resistance training
- high load frail (Experimental): Frail participants who will receive resistance training at 70% of their maximal strength
  Interventions: Other: resistance training
- low load frail (Experimental): Frail participants who will receive resistance training at 30% of their maximal strength
  Interventions: Other: resistance training

INTERVENTIONS:
Other: resistance training — Moving muscles against loads with the purpose of increasing strength.

SUMMARY:
After the age of 40-45 years muscle mass and function progressively decline, reducing older peoples' abilities to perform tasks of daily living and also increase the risk of falls. It is known that, across the life course, resistance exercise can be of benefit in increasing muscle mass and function, yet how hard the exercise should be performed has received little attention. Current recommendations are for older people to perform exercise at 70% of the maximum they can lift, quite a high intensity that often puts older people off participating. Recent evidence in younger people has suggested that such intensities are not required.

The investigators aim to determine the feasibility of a study to investigate recruitment and adherence of older people to a study of exercise training at different intensities.

DETAILED DESCRIPTION:
The cohort will comprise two sets of participants: frail older adults and non-frail older adults.

Each participant will receive 8 weeks of twice weekly supervised resistance training. Both the frail and non-frail participants will be randomised into either receiving high load resistance training or low load resistance training. High load resistance training will be delivered at 70% of the participants maximal capacity and low load resistance training will be delivered at 30% of maximal capacity. All resistance training will focus on the lower limb and regardless of intensity each exercise will be done to failure (unable to complete another full repetition).

ELIGIBILITY:
Inclusion Criteria:

Non-frail - Over 65 years of age Frail - Over 65 years of age, Three or more of the following criteria: >10lbs of weight loss unintentionally in previous year; grip strength in lowest 20% (by sex and BMI); self-reported exhaustion; walking time for 15 feet in slowest 20% (by sex and height); physical activity in the lowest 20%.

Exclusion Criteria:

Non-frail - Current participation in an exercise programme. Clinical team do not think resistance exercise would be safe or unable to consent. Any other reason that precludes participation in exercise, decision made by research team in consultation with a consultant in Geriatric Medicine where required.

Frail - Current participation in an exercise programme. Clinical team do not think resistance exercise would be safe or unable to consent. Any other reason that precludes participation in exercise, decision made by research team in consultation with a consultant in Geriatric Medicine where required.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-21 (Actual); Primary Completion 2019-11-29 (Estimated); Study Completion 2019-11-29 (Estimated)

PRIMARY OUTCOMES:
Number of training sessions attended | 8 weeks
  Expressed as a percentage of number of sessions attended
Compliance with protocol | 8 weeks
  Expressed as a percentage of number of sessions where training protocol was adhered to
Number of treatment-related adverse events as assessed by CTCAE v4.0 | 8 weeks
  Number of adverse events that could be attributed to the intervention
Acceptability of intervention (qualitative) | 8 weeks
  focus groups with semi-structured discussion plans will investigate the acceptability of the intervention

SECONDARY OUTCOMES:
Muscle thickness | 8 weeks
  Thickness of vastus lateralus using ultrasound (mm)
Muscle power | 8 weeks
  Maximum voluntary contraction of a muscle at a set angle to produce a torque (kg)
Muscle strength | 8 weeks
  Maximal load participant can lift (kg)
Frailty | 8 weeks
  As measured by the Fried criteria. These are low energy expenditure, slow gait speed, weak grip strength, exhaustion, and unintentional weight loss. Fulfilling three of these criteria indicates clinical frailty.
Quality of life | 8 weeks
  Measured using the Euroqol EQ-5 Dimension- 5 Level self report measure. This scale measures quality of life in 5 dimensions and produces an index of quality of life rangin from a worst quality of life at -1 to best quality of life at 1.
Activities of daily living | 8 weeks
  Measured using the Barthel index. This scale measures ten variables of activities of daily living and produces an overall score. This ranges from 0-20 with a higher score indicating greater independence.
Activities of daily living | 8 weeks
  Measured using the Lawton ADL scale. this self report measures assess independence in daily living in 8 different domains but produces an overall score. Scores range from 0-8 with 8 indicating full independence.
Functional abilities | 8 weeks
  Short performance battery test. This battery of tests assesses balance, gait speed and lower limb strength. Scores are awarded for each individual section and aggregated ranging from 0-12 with a higher score indicating greater physical capability.
motion analysis | 8 weeks
  biomechanical assessment using infr-red motion analysis cameras

CONTACTS AND LOCATIONS:
Overall Officials: Evan Campbell, PhD, Principal Investigator — Univeristy of Glasgow
Locations (1):
- Glasgow Royal Infirmary, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No